CLINICAL TRIAL: NCT00160537
Title: A Monocenter, Double-blind, Randomized Trial, With Two Parallel Groups Comparing the Clinical Efficacy of Levocetirizine 5 mg Capsules and Desloratadine 5 mg Capsules Taken Once a Day Over 3 Weeks of Treatment in Adult Subjects Suffering From Seasonal Allergic Rhinitis (SAR) Due to Grass Pollen
Brief Title: POPULAR (Preference Of Patient Using Levocetirizine in Allergic Rhinitis)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: A00391; EudraCT 2004-002971-18; POPULAR
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2009-09

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Seasonal Allergic Rhinitis (SAR), Grass pollen, SAR Symptoms (sneezing, rhinorrhea, nasal / ocular pruritus, nasal congestion); POPULAR, Xyzal, Levocetirizine
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Sneezing; Rhinorrhea; Nasal Obstruction | interventions — levocetirizine

INTERVENTIONS:
Drug: Levocetirizine

SUMMARY:
Comparative study on clinical efficacy and safety of levocetirizine and desloratadine as measured by the subject's satisfaction/dissatisfaction after one week of treatment

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of SAR known and treated since 2 years.
* Positive skin prick test (wheal > 3 mm larger than the diluent control) or RAST (≥3.5 IU/ml) to grass pollen (less than 1 year).
* Minimum mean T5SS of 8 during the baseline period.

Exclusion Criteria:

* Have an associated asthma requiring a daily treatment other than β2 short acting agonist prn
* Have atopic dermatitis or urticaria requiring antihistamine treatment or the administration of oral or topical corticosteroids and any other disease requiring the administration of oral or topical corticosteroids

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-05; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Subjects' satisfaction / dissatisfaction after the first week of treatment.

SECONDARY OUTCOMES:
allergic rhinitis symptoms scores over the first week of treatment , subject's satisfaction / dissatisfaction of their choice of treatment after the first week of treatment, time to first feeling of (sufficient) symptom improvement during the first we

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma